CLINICAL TRIAL: NCT06263816
Title: Effect of Long-term Carvedilol to Prevent Decompensation or Death in Patients With Asymptomatic Child-Pugh A5 to B8 Cirrhosis and Clinically Significant Portal Hypertension: a Multicenter Double-blind Randomized Control Trial
Acronym: CARVECIR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Centre Hospitalier Universitaire Amiens Picardie (Unknown); Centre Hospitalier Universitaire Angers (Unknown); Assistance Publique Hopitaux Paris BEAUJON (Unknown); Centre Hospitalier Universitaire Caen (Unknown); Centre Hospitalier intercommunal de Créteil (Unknown); Hospices Civils de Lyon (Other); Centre Hospitalier Universitaire Grenoble (Unknown); Centre Hospitalier Universitaire Haut Lévêque (Unknown); Centre Hospitalier Régional Universitaire Lille (Unknown); Centre Hospitalier Universitaire Jean Minjoz (Unknown); Assistance Publique Hopitaux Paris AVICENNE (Unknown); Centre Hospitalier Universitaire Clermont Ferrand (Unknown); Assistance Publique Hopitaux Paris LA PITIE SALPETRIERE (Unknown); Centre Hospitalier Universitaire Pontchaillou (Unknown); Assistance Publique Hopitaux Paris ST ANTOINE (Unknown); Assistance Publique Hopitaux Paris PAUL BROUSSE (Unknown); University Hospital, Montpellier (Other); Assistance Publique Hopitaux Paris HENRI MONDOR (Unknown); Centre Hospitaliser Départemental de Vendée (Unknown); Nantes University Hospital (Other); Centre Hospitalier Universitaire Dijon (Other); CHU de Reims (Other); Hôpitaux Universitaires de Strasbourg (Unknown); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CARVECIR
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Asymptomatic Cirrhosis; Clinically Significant Portal Hypertension
Keywords: carvedilol; decompensation; death; asymptomatic cirrhosis; significant portal hypertension
MeSH Terms: conditions — Death | interventions — Carvedilol

STUDY DESIGN:
Intervention Model Description: This study will be a national multicentric, phase III, superiority double-blinded randomized controlled trial with two parallel arms: carvedilol versus placebo. The primary end-point will be assessed by the local investigator (hepatologist), blinded of the randomization arm
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carvédilol (Experimental)
  Interventions: Drug: Experimental group: Patients will be treated with carvedilol.
- Placebo (Placebo Comparator)
  Interventions: Other: Control group: Patients will receive a placebo.

INTERVENTIONS:
Drug: Experimental group: Patients will be treated with carvedilol. — Patients will receive the number of pills of carvedilol corresponding to the dose determined during the titration period (either one pill of 6.25 mg in the morning or 1 pill of 6.25 mg twice a day, 1 in the morning and 1 in the evening.
  Arms: Carvédilol
Other: Control group: Patients will receive a placebo. — Patients will receive the number of pills of placebo corresponding to the dose determined during the titration period (either one pill in the morning or 1 pill twice a day: 1 in the morning and 1 in the evening).
  Arms: Placebo

SUMMARY:
Decompensation of cirrhosis is a turning point in cirrhosis course, as associated with a marked decrease in life expectancy. Thus, prevention of decompensation is crucial.

The usefulness of carvedilol to prevent decompensation of cirrhosis in patients with TE-LSM ≥ 25 kPa as a surrogate marker for clinically significant portal hypertension, has never been evaluated in a clinical trial.

DETAILED DESCRIPTION:
Decompensation of cirrhosis is a turning point in cirrhosis course, as associated with a marked decrease in life expectancy. Thus, prevention of decompensation is crucial.

Portal hypertension (PH) is the strongest predictor of decompensation. Hepatic venous pressure gradient (HVPG) is the reference standard for the evaluation of PH. HVPG ≥10 mm Hg, called "clinically significant portal hypertension", identifies a population with a high risk of decompensation. HVPG measurement is an invasive procedure, only routinely available in expert centers. Liver stiffness measurement (LSM) using transient elastography (TE) (referred as TE LSM) using Fibroscan can provide an indirect estimate of HVPG. TE-LSM ≥ 25 kPa can rule-in HVPG ≥10 mm Hg with a specificity >90%.

Nonselective beta-blockers (NSBBs) lower portal pressure by decreasing portal venous inflow. Carvedilol also decreases intrahepatic vascular resistance, and thereby achieves a greater reduction in portal pressure than propranolol. At low-dose (≤12.5 mg/day), carvedilol is safe in patients with compensated cirrhosis.

In patients with asymptomatic cirrhosis, NSBBs were recommended when medium or large varices (high-risk varices) are present for prophylaxis of variceal bleeding. In a recent randomized controlled trial, the PREDESCI study (NCT01059396), NSBBs reduced incidence of decompensation or death in patients with compensated cirrhosis with clinically significant portal hypertension. In the PREDESCI study, the diagnosis of clinically significant portal hypertension was based on invasive HVPG measurement, so that its results are not applicable in clinical practice.

The usefulness of carvedilol to prevent decompensation of cirrhosis in patients with TE-LSM ≥25 kPa as a surrogate marker for clinically significant portal hypertension, has never been evaluated in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female≥ 18 years of age
* Cirrhosis related to hepatitis C or hepatitis B virus without viral replication for at least 2 years.

Or Cirrhosis related to alcohol consumption (active or abstinent) Or Cirrhosis related to metabolic syndrome or cryptogenic with BMI < 30 kg/m2

* 2 TE-LSM (Fibroscan®) performed in fasting conditions, using either the M or the XL probe >=25 kPa, within 12 months before inclusion
* Absence of medium or large varices or small varices with red signs at endoscopy within 3 months before inclusion
* Child-Pugh A5 to B8
* Affiliation to a French social security system.
* Written informed consent obtained from the participant or participant's legal representative
* For child-bearing aged women, contraception using oral contraceptive, or intrauterine device or mechanical contraception

Exclusion Criteria:

* History of overt ascites or encephalopathy <12 months before inclusion
* Treatment with either diuretics or lactulose or rifaximin <3 months before inclusion
* Any history of portal hypertension related bleeding
* Baseline heart rate <65/min or systolic blood pressure <100 mm Hg
* Previous transjugular intrahepatic portosystemic shunt (TIPSS) or liver transplantation
* Previous history or active hepatocellular carcinoma
* Glomerular filtration rate (CKD-Epi) < 30 mL/min
* Strict indication to selective or nonselective beta-blockers: history of acute myocardial infarction, congestive heart failure
* Strict contraindication to selective or nonselective beta-blockers:

  * decompensated congestive heart failure
  * grade 2 or 3 atrioventricular block
  * sinus node dysfunction without pacemaker
  * severe asthma according to WHO classification [63]
  * severe Chronic Obstructive Pulmonary Disease, defined stage 3 or 4 of the GOLD classification, i.e.FEV1<50% of the predicted value (https://goldcopd.org/)
  * severe Raynaud disease, defined as repetitive episodes of biphasic colour (at least two) of pallor, cyanosis, erythema, in addition to paresthesia or numbness, occurring in both cold and normal environments [64].
* Known hypersensitivity to carvedilol
* Concomitant use of Cimétidin
* Concomitant use of class I antiarythmic agents (except lidocaïn) (i.e.cibenzoline, disopyramide, flécaïnide, hydroquinidine méxilétine, propafenone, quinidine)
* Concomitant use of calcium antagonists: diltiazem, vérapamil and bépridil
* Concomitant use of clonidine, méthyldopa, guanfacine, moxonidine, rilménidine
* Concomitant use of fingolimod
* Concomitant use of potent inhibitors (e.g. ketoconazole, HIV protease inhibitors) or inductors (e.g. rifampin, carbamazepine, phenytoin) of CYP3A4 (see appendix 7)
* Pregnancy or breastfeeding
* Non ability for participant to comply with the requirements of the study
* Life expectancy <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-06-17 (Estimated); Primary Completion 2027-07-17 (Estimated); Study Completion 2030-07-17 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of low dose carvedilol (<=12.5 mg per day) versus placebo on the occurrence of decompensation of cirrhosis or liver-related death at 36 months | 36 months
  Primary endpoint will be the occurrence, within 36 months after inclusion, of either decompensation of cirrhosis or liver-related death.
  Decompensation of cirrhosis is defined as a composite endpoint including one event among: overt ascites, overt hepatic encephalopathy and variceal bleeding according to Baveno VII consensus conference [1].
  Liver-related death is defined as death occurring in the context of complicated ascites (e.g. spontaneous bacterial peritonitis or acute kidney injury), encephalopathy, variceal hemorrhage, or ACLF

CONTACTS AND LOCATIONS:
Overall Officials: Laure ELKRIEF, MD-PhD, Study Director — University Hospital, Tours
Locations (24):
- France (24):
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - CHU Beaujon, Assistance Publique Hôpitaux de Paris
  - CHU Jean Minjoz, Besançon
  - CHU Haut Lévêque, Bordeaux
  - CHU Caen, Caen
  - CH intercommunal de Créteil, CH Intercommunal de Créteil
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Hôpital Francois Mitterrand, Dijon
  - CHU Grenoble, Grenoble
  - Centre Hospitalier départemental de Vendée, La Roche-sur-Yon
  - Hôpital Huriez, Lille
  - CHU la Croix Rousse, Lyon
  - CHU de Montpellier, Montpellier
  - CHU Hôtel Dieu, Nantes
  - CHU Avicenne, Paris
  - CHU Pitié-Salpêtrière, Paris
  - CHU Saint-Antoin, Paris
  - CHU de Reims, Reims
  - CHU Pontchaillou, Rennes
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No